CLINICAL TRIAL: NCT01727297
Title: REVEAL AF: Incidence of AF in High Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: REVEAL AF
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- REVEAL Implantable Cardiac Monitor (Other)
  Interventions: Device: REVEAL Implantable Cardiac Monitor

INTERVENTIONS:
Device: REVEAL Implantable Cardiac Monitor

SUMMARY:
This study is to determine, through continuous monitoring with the Reveal implantable cardiac monitor (ICM), the incidence of atrial fibrillation (AF) in patients suspected to be at high risk for having AF and to understand how physicians manage these patients after AF has been detected. This study will also seek to identify what patient characteristics are most predictive of developing AF.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets the approved indications to receive the Reveal ICM
* Patient is suspected, based on symptomatology and/or demographics, of having atrial fibrillation or at high risk of having AF, as determined by the clinical investigator
* Patient has a Congestive heart failure, Hypertension, Age ≥75 years, Diabetes mellitus, prior Stroke or transient ischemic attack (TIA) or thromboembolism (doubled) (CHADS2) score ≥ 3 OR has a CHADS2 score = 2 with at least one of the following documented: renal impairment (GFR 30-60 ml/min), sleep apnea, coronary artery disease, or chronic obstructive pulmonary disease. Note: stroke/TIA criterion as part of the CHADS2 score for this trial is limited to either an ischemic stroke or TIA, which occurred more than one year prior to enrollment.
* Patient is 18 years of age or older
* Patient has a life expectancy of 18 months or more
* Patient, or legally authorized representative, is willing to sign and date the consent form
* Patient is willing and able to be remotely monitored (i.e., eligible for enrollment into the Medtronic CareLink Network)

Exclusion Criteria:

* Patient has a documented history of AF or atrial flutter
* Patient had an ischemic stroke or TIA within past year prior to enrollment
* Patient has a history of a hemorrhagic stroke
* Patient is currently implanted with an implantable pulse generator (IPG), implantable cardioverter defibrillator (ICD), cardiac resynchronization therapy pacemaker (CRT-P), or cardiac resynchronization therapy defibrillator (CRT-D) device
* New York Heart Association (NYHA) Class IV Heart Failure patient
* Patient had heart surgery within previous 90 days prior to enrollment
* Patient had a myocardial infarction (MI) within the previous 90 days prior to enrollment
* Patient is taking chronic immuno-suppressant therapy
* Patient is taking an anti-arrhythmic drug
* Patient is contraindicated for long term anticoagulation medication
* Patient is taking a long-term anticoagulation medication
* Any concomitant condition which, in the opinion of the investigator, would not allow safe participation in the study (e.g., drug addiction, alcohol abuse, emotional / psychological diagnosis)
* Patient is enrolled in another study that could confound the results of this study, without documented pre-approval from Medtronic study manager
* Patient has a creatinine clearance <30 ml/min or is on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2012-11-13 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Reiffel, MD, Principal Investigator — Columbia University
Locations (58):
- United States (43):
  - Phoenix Heart, PLLC, Glendale, Arizona
  - Cardiovascular Consultants Heart Center, Fresno, California
  - Desert Heart Rhythm Consultants, Palm Springs, California
  - Healdsburg Cardiology, Windsor, California
  - Nanticoke Cardiology, Seaford, Delaware
  - Bradenton Cardiology, Bradenton, Florida
  - The Cardiac & Vascular Institute, Gainesville, Florida
  - Cardiac Clinic, Kissimmee, Florida
  - Northside Hospital, St. Petersburg, Florida
  - North Georgia Heart Foundation, Gainesville, Georgia
  - Premier HealthCare, Bloomington, Indiana
  - Cardiovascular Consultants PC (Munster IN), Munster, Indiana
  - The University Kansas Medical Center Research Institute Inc, Kansas City, Kansas
  - Cardiovascular Consultants of Kansas, Wichita, Kansas
  - Delmarva Heart Research Foundation Inc, Salisbury, Maryland
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Cox Medical Center South, Springfield, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Glacier View Research Institute Cardiology, Kalispell, Montana
  - CHI Health Cardiology (Bergen), Omaha, Nebraska
  - Englewood Hospital & Medical Center, Englewood, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - New York-Presbyterian Hospital/Columbia University Medical Center, New York, New York
  - Caromont Regional Medical Center, Gastonia, North Carolina
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - Salem Cardiovascular Associates, Salem, Oregon
  - The Heart Care Group PC (Allentown PA), Allentown, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - South County Cardiology, Wakefield, Rhode Island
  - Selcuk A. Tombul, D.O., F.A.C.C., Chattanooga, Tennessee
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - Sutherland Cardiology Clinic, Germantown, Tennessee
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - Baylor Research Institute (Plano TX), Plano, Texas
  - Woodlands North Houston Heart and Vein Center, The Woodlands, Texas
  - ProHealth Care, Waukesha, Wisconsin
- Austria (2):
  - LKH - Universitätsklinikum Graz, Graz
  - Allgemein öffentliches Krankenhaus der Elisabethinen Linz, Linz
- Germany (6):
  - Klinikum Coburg GmbH, Coburg
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsmedizin Göttingen Georg-August-Universität, Göttingen
  - Asklepios Klinik Sankt Georg, Hamburg
  - Klinikum Lünen St.-Marien-Hospital GmbH - Akademisches Lehrkrankenhaus der Westfälischen Wilhelms-Un, Lünen
  - Eberhard Karls Universität Tübingen - Universitätsklinikum Tübingen, Tübingen
- Italy (3):
  - Azienda Ospedaliera San Gerardo, Monza
  - Ospedale classificato ed equiparato Sacro Cuore - Don Calabria, Negrar
  - Ospedale civile di Ciriè, Torino
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - St. Antonius Ziekenhuis, Nieuwegein
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Hospital Universitari de Tarragona Joan XXIII, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reiffel JA, Verma A, Kowey PR, Halperin JL, Gersh BJ, Elkind MSV, Ziegler PD, Kaplon RE, Sherfesee L, Wachter R; REVEAL AF Investigators. Rhythm monitoring strategies in patients at high risk for atrial fibrillation and stroke: A comparative analysis from the REVEAL AF study. Am Heart J. 2020 Jan;219:128-136. doi: 10.1016/j.ahj.2019.07.016. PMID 31862084
- [Derived] Reiffel JA, Verma A, Kowey PR, Halperin JL, Gersh BJ, Wachter R, Pouliot E, Ziegler PD; REVEAL AF Investigators. Incidence of Previously Undiagnosed Atrial Fibrillation Using Insertable Cardiac Monitors in a High-Risk Population: The REVEAL AF Study. JAMA Cardiol. 2017 Oct 1;2(10):1120-1127. doi: 10.1001/jamacardio.2017.3180. PMID 28842973

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients in the 'No Reveal Implantable Cardiac Monitor Implant Attempt' arm were exited from the study prior to an implant attempt. Therefore, no outcome data are available. Baseline data are not presented due to variable data collection before the time of exit. Adverse event data were collected for this cohort, and are reported below.
Groups:
- Reveal Implantable Cardiac Monitor Implant Attempted: Enrolled subjects who had a Reveal Implantable Cardiac Monitor implant attempt (i.e. underwent the procedure to have a Reveal device implanted)
- No Reveal Implantable Cardiac Monitor Implant Attempt: Enrolled subjects who exited the study prior to undergoing a procedure to implant a Reveal Implantable Cardiac Monitor
Period: Overall Study
Arm/Group | Reveal Implantable Cardiac Monitor Implant Attempted | No Reveal Implantable Cardiac Monitor Implant Attempt
Started | 395 | 51
Completed | 293 | 0
Not Completed | 102 | 51
Not completed — Death | 13 | 0
Not completed — Protocol Violation | 1 | 10
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 11 | 0
Not completed — Withdrawal by Subject | 26 | 27
Not completed — Physician Decision | 19 | 5
Not completed — Other (e.g. AF detection pre-implant) | 29 | 8

BASELINE CHARACTERISTICS:
Arm/Group | Reveal Implantable Cardiac Monitor Implant Attempted
Number analyzed (Participants) | 395
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 88
  >=65 years | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188
  Male | 207
Region of Enrollment [Number; unit: participants]
  Austria | 18
  Netherlands | 6
  United States | 302
  Italy | 19
  Slovenia | 4
  Germany | 39
  Spain | 7

OUTCOME MEASURES:

1. Primary Outcome: 18 Month Incidence Rate of Atrial Fibrillation (AF) Lasting Six or More Minutes
Description: Incidence of adjudicated AF lasting six or more minutes at 18 months. Each arrhythmic episode detected by the patient's Reveal device will be reviewed to determine if it is 1) an actual atrial fibrillation episode, and (2) is at least 6 minutes in duration. The first such episode per patient occurring within 18 months will be utilized to determine the 18 month incidence rate.
Time Frame: Implant to 18 months post device insertion
Population: This analysis only included patients who received an implantable cardiac monitor, met all inclusion/exclusion criteria, and had device data available. Of the 395 participants who underwent an implant attempt, 1 attempt was unsuccessful, 7 subjects did not meet all inclusion/exclusion criteria, and 2 subjects had no post-implant device data.
Measure: Number; unit: percent of participants
Groups:
- Primary Objective Analysis Cohort: Subjects successfully implanted with a Reveal Implantable Cardiac Monitor (ICM), who also (1) have post-implant device data to evaluate, (2) were not on anti-arrhythmic medication at enrollment, (3) did not have AF prior to Reveal ICM implant, and (4) satisfy the Congestive heart failure, Hypertension, Age ≥75 years, Diabetes mellitus, prior Stroke or transient ischemic attack (TIA) or thromboembolism (doubled) (CHADS2) inclusion criteria for the study (CHADS2 score of 3 or higher, or a CHADS2 score of 2 along with chronic obstructive pulmonary disease, sleep apnea, renal impairment, or coronary artery disease)
Arm/Group | Primary Objective Analysis Cohort
Number analyzed (Participants) | 385
percent of participants | 29.3

2. Secondary Outcome: Predictors of the Incidence of AF
Description: AF will be defined as in the primary outcome. Baseline characteristics including demographics, medical history, and biomarkers at enrollment will be tested for their association with a patient's risk of developing AF.
Time Frame: Time from implant to date of last stored available device data (maximum of 30 months)
Population: This analysis only included patients who received an implantable cardiac monitor, were not on antiarrhythmic medications at baseline, and had device data available. Of the 395 participants who underwent an implant attempt, 1 attempt was unsuccessful, 1 subject was on antiarrhythmic medication, and 2 subjects had no post-implant device data.
Measure: Count of Participants; unit: Participants
Groups:
- AF Predictors Analysis Cohort: AF Episodes: Subjects successfully implanted with a Reveal Implantable Cardiac Monitor (ICM), and who (1) have post-implant ICM device data to evaluate, (2) were not on anti-arrhythmic medication at enrollment, (3) did not have AF prior to Reveal implant, and (4) experienced an AF episode lasting at least 6 minutes during follow-up.
- AF Predictors Analysis Cohort: No AF Episodes: Subjects successfully implanted with a Reveal Implantable Cardiac Monitor (ICM), and who (1) have post-implant ICM device data to evaluate, (2) were not on anti-arrhythmic medication at enrollment, (3) did not have AF prior to Reveal implant, and (4) did not experience an AF episode lasting at least 6 minutes during follow-up.
Arm/Group | AF Predictors Analysis Cohort: AF Episodes | AF Predictors Analysis Cohort: No AF Episodes
Number analyzed (Participants) | 130 | 261
Participants
  Gender (Male) | 67 | 138
  Diabetes | 80 | 168
  Heart failure | 31 | 50
  Hypertension | 122 | 244
  Renal impairment | 60 | 106
  Chronic obstructive pulmonary disorder | 19 | 57
  Prior stroke > 1 year ago | 23 | 56
  Coronary artery disease | 75 | 157
  Sleep apnea | 28 | 75
  Family history of AF | 5 | 3
  Vascular disease | 25 | 54
Statistical Analysis 1: Comparison: AF Predictors Analysis Cohort: AF Episodes vs AF Predictors Analysis Cohort: No AF Episodes; The null hypothesis was that age did not influence a patient's risk of experiencing AF (it's coefficient in a Cox proportional hazards model was 0); Test type: Superiority; p < 0.001, Regression, Cox — All predictors were tested in a multivariable Cox proportional hazards regression model; the results were not adjusted for multiple comparisons. Age was treated as a continuous variable in years; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [1.05 to 1.11] — The hazard ratio represented the effect of a one year increase in age on a patient's risk of developing AF. Descriptive statistics (mean±standard deviation) for age were 75.7±7.9 years among patients with AF, and 69.4±10.0 among patients without AF
Statistical Analysis 2: Comparison: AF Predictors Analysis Cohort: AF Episodes vs AF Predictors Analysis Cohort: No AF Episodes; The null hypothesis was that body mass index (BMI) did not influence a patient's risk of experiencing AF (it's coefficient in a Cox proportional hazards model was 0); Test type: Superiority; p = 0.02, Regression, Cox — All predictors were tested in a multivariable Cox proportional hazards regression model; the results were not adjusted for multiple comparisons. BMI was treated as a continuous variable; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [1.01 to 1.08] — The hazard ratio represented the effect of a one unit increase in BMI on a patient's risk of developing AF. Descriptive statistics (mean ± standard deviation) for BMI were 31.0 ± 6.6 among patients with AF, and 31.2 ± 6.4 among patients without AF
Statistical Analysis 3: Comparison: AF Predictors Analysis Cohort: AF Episodes vs AF Predictors Analysis Cohort: No AF Episodes; The null hypothesis was that gender did not influence a patient's risk of experiencing AF (it's coefficient for being male in a Cox proportional hazards model was 0); Test type: Superiority; p = 0.56, Regression, Cox — All predictors were tested in a multivariable Cox proportional hazards regression model; the results were not adjusted for multiple comparisons; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.77 to 1.61] — The hazard ratio represented the effect of being male on a patient's risk of developing AF
Statistical Analysis 4: Comparison: AF Predictors Analysis Cohort: AF Episodes vs AF Predictors Analysis Cohort: No AF Episodes; The null hypothesis was that diabetes did not influence a patient's risk of experiencing AF (it's coefficient in a Cox proportional hazards model was 0); Test type: Superiority; p = 0.66, Regression, Cox — [p-value comment as in outcome 2, analysis 3]; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.74 to 1.59] — The hazard ratio represented the effect of having diabetes on a patient's risk of developing AF
Statistical Analysis 5: Comparison: AF Predictors Analysis Cohort: AF Episodes vs AF Predictors Analysis Cohort: No AF Episodes; The null hypothesis was that heart failure did not influence a patient's risk of experiencing AF (it's coefficient in a Cox proportional hazards model was 0); Test type: Superiority; p = 0.73, Regression, Cox — [p-value comment as in outcome 2, analysis 3]; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.69 to 1.69] — The hazard ratio represented the effect of having heart failure on a patient's risk of developing AF
Statistical Analysis 6: Comparison: AF Predictors Analysis Cohort: AF Episodes vs AF Predictors Analysis Cohort: No AF Episodes; The null hypothesis was that hypertension did not influence a patient's risk of experiencing AF (it's coefficient in a Cox proportional hazards model was 0); Test type: Superiority; p = 0.58, Regression, Cox — [p-value comment as in outcome 2, analysis 3]; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.58 to 2.60] — The hazard ratio represented the effect of having hypertension on a patient's risk of developing AF
Statistical Analysis 7: Comparison: AF Predictors Analysis Cohort: AF Episodes vs AF Predictors Analysis Cohort: No AF Episodes; The null hypothesis was that renal impairment did not influence a patient's risk of experiencing AF (it's coefficient in a Cox proportional hazards model was 0); Test type: Superiority; p = 0.65, Regression, Cox — [p-value comment as in outcome 2, analysis 3]; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.64 to 1.32] — The hazard ratio represented the effect of having renal impairment on a patient's risk of developing AF
Statistical Analysis 8: Comparison: AF Predictors Analysis Cohort: AF Episodes vs AF Predictors Analysis Cohort: No AF Episodes; The null hypothesis was that Chronic obstructive pulmonary disease (COPD) did not influence a patient's risk of experiencing AF (it's coefficient in a Cox proportional hazards model was 0); Test type: Superiority; p = 0.22, Regression, Cox — [p-value comment as in outcome 2, analysis 3]; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.45 to 1.20] — The hazard ratio represented the effect of having COPD on a patient's risk of developing AF
Statistical Analysis 9: Comparison: AF Predictors Analysis Cohort: AF Episodes vs AF Predictors Analysis Cohort: No AF Episodes; The null hypothesis was that prior stroke more than one year pre-device implant did not influence a patient's risk of experiencing AF (it's coefficient in a Cox proportional hazards model was 0); Test type: Superiority; p = 0.53, Regression, Cox — [p-value comment as in outcome 2, analysis 3]; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.54 to 1.38] — The hazard ratio represented the effect of having a prior stroke (more than one year pre-device implant) on a patient's risk of developing AF
Statistical Analysis 10: Comparison: AF Predictors Analysis Cohort: AF Episodes vs AF Predictors Analysis Cohort: No AF Episodes; The null hypothesis was that coronary artery disease did not influence a patient's risk of experiencing AF (it's coefficient in a Cox proportional hazards model was 0); Test type: Superiority; p = 0.21, Regression, Cox — [p-value comment as in outcome 2, analysis 3]; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.53 to 1.15] — The hazard ratio represented the effect of having coronary artery disease on a patient's risk of developing AF
Statistical Analysis 11: Comparison: AF Predictors Analysis Cohort: AF Episodes vs AF Predictors Analysis Cohort: No AF Episodes; The null hypothesis was that sleep apnea did not influence a patient's risk of experiencing AF (it's coefficient in a Cox proportional hazards model was 0); Test type: Superiority; p = 0.19, Regression, Cox — [p-value comment as in outcome 2, analysis 3]; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.45 to 1.17] — The hazard ratio represented the effect of having sleep apnea on a patient's risk of developing AF
Statistical Analysis 12: Comparison: AF Predictors Analysis Cohort: AF Episodes vs AF Predictors Analysis Cohort: No AF Episodes; The null hypothesis was that family history of AF did not influence a patient's risk of experiencing AF (it's coefficient in a Cox proportional hazards model was 0); Test type: Superiority; p = 0.16, Regression, Cox — [p-value comment as in outcome 2, analysis 3]; Hazard Ratio (HR) = 1.97, 95% CI 2-sided [0.76 to 5.14] — The hazard ratio represented the effect of having a family history of AF on a patient's risk of developing AF
Statistical Analysis 13: Comparison: AF Predictors Analysis Cohort: AF Episodes vs AF Predictors Analysis Cohort: No AF Episodes; The null hypothesis was that vascular disease did not influence a patient's risk of experiencing AF (it's coefficient in a Cox proportional hazards model was 0); Test type: Superiority; p = 0.63, Regression, Cox — [p-value comment as in outcome 2, analysis 3]; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.56 to 1.43] — The hazard ratio represented the effect of having vascular disease on a patient's risk of developing AF

3. Secondary Outcome: Actions Taken in Response to Awareness of AF
Description: Clinical actions taken in response to clinician awareness of a patient's AF onset or progression will be summarized
Time Frame: Time from first identified episode of AF to study exit (maximum of 30 months)
Population: Each visit represents the number of subjects who had a 1st, 2nd, 3rd visit, etc. in which AF was identified by the physician. Subjects in the "Sixth Visit with AF Detected" column had 6 visits in which AF was detected by the physician, and the column reflects the actions taken at that sixth visit.
Measure: Count of Units; unit: Actions at Visits
Units Other Than Participants: Actions at Visits
Groups:
- First Visit With AF Detected: Enrolled subjects implanted with a Reveal Implantable Cardiac Monitor who:
  1. Did not have diagnosed AF prior to implant,
  2. met the CHADS2 score inclusion criterion (a CHADS2 score of at least 3 or a CHADS2 score of 2 with at least one of the following: coronary artery disease, sleep apnea, renal impairment, or chronic obstructive pulmonary disease),
  3. was not taking an anti-arrhythmic drug at enrollment, and
  4. Had a follow-up visit in which new AF episodes were diagnosed
- Second Visit With AF Detected: Enrolled subjects implanted with a Reveal Implantable Cardiac Monitor who:
  1. Did not have diagnosed AF prior to implant,
  2. met the CHADS2 score inclusion criterion (a CHADS2 score of at least 3 or a CHADS2 score of 2 with at least one of the following: coronary artery disease, sleep apnea, renal impairment, or chronic obstructive pulmonary disease),
  3. was not taking an anti-arrhythmic drug at enrollment, and
  4. Had a 2nd follow-up visit in which new AF episodes were diagnosed
- Third Visit With AF Detected: Enrolled subjects implanted with a Reveal Implantable Cardiac Monitor who:
  1. Did not have diagnosed AF prior to implant,
  2. met the CHADS2 score inclusion criterion (a CHADS2 score of at least 3 or a CHADS2 score of 2 with at least one of the following: coronary artery disease, sleep apnea, renal impairment, or chronic obstructive pulmonary disease),
  3. was not taking an anti-arrhythmic drug at enrollment, and
  4. Had a 3rd follow-up visit in which new AF episodes were diagnosed
- Fourth Visit With AF Detected: Enrolled subjects implanted with a Reveal Implantable Cardiac Monitor who:
  1. Did not have diagnosed AF prior to implant,
  2. met the CHADS2 score inclusion criterion (a CHADS2 score of at least 3 or a CHADS2 score of 2 with at least one of the following: coronary artery disease, sleep apnea, renal impairment, or chronic obstructive pulmonary disease),
  3. was not taking an anti-arrhythmic drug at enrollment, and
  4. Had a 4th follow-up visit in which new AF episodes were diagnosed
- Fifth Visit With AF Detected: Enrolled subjects implanted with a Reveal Implantable Cardiac Monitor who:
  1. Did not have diagnosed AF prior to implant,
  2. met the CHADS2 score inclusion criterion (a CHADS2 score of at least 3 or a CHADS2 score of 2 with at least one of the following: coronary artery disease, sleep apnea, renal impairment, or chronic obstructive pulmonary disease),
  3. was not taking an anti-arrhythmic drug at enrollment, and
  4. Had a 5th follow-up visit in which new AF episodes were diagnosed
- Sixth Visit With AF Detected: Enrolled subjects implanted with a Reveal Implantable Cardiac Monitor who:
  1. Did not have diagnosed AF prior to implant,
  2. met the CHADS2 score inclusion criterion (a CHADS2 score of at least 3 or a CHADS2 score of 2 with at least one of the following: coronary artery disease, sleep apnea, renal impairment, or chronic obstructive pulmonary disease),
  3. was not taking an anti-arrhythmic drug at enrollment, and
  4. Had a 6th follow-up visit in which new AF episodes were diagnosed
Arm/Group | First Visit With AF Detected | Second Visit With AF Detected | Third Visit With AF Detected | Fourth Visit With AF Detected | Fifth Visit With AF Detected | Sixth Visit With AF Detected
Number analyzed (Participants) | 115 | 57 | 31 | 20 | 12 | 6
Number analyzed (Actions at Visits) | 85 | 14 | 6 | 4 | 2 | 0
Actions at Visits
  Oral Anticoagulation Initiated | 61 | 5 | 0 | 1 | 2 | 0
  Rhythm Control Medication Initiated | 13 | 2 | 0 | 1 | 0 | 0
  Rate Control Medication Initiated | 4 | 3 | 2 | 1 | 0 | 0
  Cardioversion | 2 | 2 | 1 | 0 | 0 | 0
  Ablation | 0 | 2 | 3 | 1 | 0 | 0
  Referral to Another Physician | 5 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events occurring from the time of enrollment (consent) until exit will be included. All subjects were to be followed a minimum of 18 months and a maximum of 30 months post-Reveal device implantation.
Arm/Group | Reveal Implantable Cardiac Monitor Implant Attempted | No Reveal Implantable Cardiac Monitor Implant Attempt
All-Cause Mortality (participants affected / at risk) | 13/395 | 0/51
Serious Adverse Events (participants affected / at risk) | 153/395 | 1/51
Other Adverse Events (participants affected / at risk) | 34/395 | 1/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reveal Implantable Cardiac Monitor Implant Attempted (N=395) | No Reveal Implantable Cardiac Monitor Implant Attempt (N=51)
Chest pain (General disorders) | 11 (15) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 10 (10) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 9 (9) | 0 (0)
Pneumonia (Infections and infestations) | 6 (8) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 8 (8) | 0 (0)
Coronary artery disease (Cardiac disorders) | 7 (7) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 5 (6) | 0 (0)
Cardiac arrest (Cardiac disorders) | 6 (6) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (6) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (6) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 6 (6) | 0 (0)
Bradycardia (Cardiac disorders) | 5 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (5) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 4 (5) | 0 (0)
Syncope (Nervous system disorders) | 5 (5) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 4 (4) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Hypertensive crisis (Vascular disorders) | 3 (4) | 0 (0)
Implant site pain (General disorders) | 4 (4) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 3 (4) | 0 (0)
Angina unstable (Cardiac disorders) | 3 (3) | 0 (0)
Asthenia (General disorders) | 3 (3) | 0 (0)
Medical device site erosion (General disorders) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Implant site infection (Infections and infestations) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Basal ganglia stroke (Nervous system disorders) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Central nervous system inflammation (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Device dislocation (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lead dislodgement (General disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Oversensing (General disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reveal Implantable Cardiac Monitor Implant Attempted (N=395) | No Reveal Implantable Cardiac Monitor Implant Attempt (N=51)
Atrial fibrillation (Cardiac disorders) | 34 (36) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, contracts allow investigators to publish study results per the protocol and publication plan. Investigators and participating institutions will provide any publication of study data generated by the Investigator and/or participating institution to Medtronic for review prior to submission to determine if confidential information ("CI") is included and to check for technical correctness. Medtronic may not censor/interfere with the publication beyond the extent necessary to protect CI.